CLINICAL TRIAL: NCT02360904
Title: A Yoga Program for Breast Cancer Patients Undergoing Chemotherapy: Effects on Quality of Life and Chemotherapy-associated Symptoms
Brief Title: A Yoga Program for Breast Cancer Patients Undergoing Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Theresa Shao, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 16-0656; 025-14 (Other: Beth Israel IRB)
Record Dates: First submitted 2015-02-06; First posted 2015-02-11 (Estimated); Last update posted 2021-08-17 (Actual); Status verified 2019-02

CONDITIONS: Fatigue; Sleep Disturbances
MeSH Terms: conditions — Fatigue; Parasomnias | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- start yoga classes immediately (Experimental): 12 weekly 60-minute yoga classes taught by a certified yoga instructor with cancer-specific yoga training that will commence concurrently with the start of chemotherapy.
  Interventions: Other: Yoga
- Start yoga classes after 3 months (Active Comparator): 12 weekly 60-minute yoga classes taught by a certified yoga instructor with cancer-specific yoga training that will commence 3 months after start of chemotherapy
  Interventions: Other: Yoga

INTERVENTIONS:
Other: Yoga — The intervention will consist of 12 weekly 60-minute yoga classes taught by a certified yoga instructor with cancer-specific yoga training. Classes will be conducted at the Beth Israel Comprehensive Cancer Center in a closed-group format, and will be offered twice a week. Yoga mats will be provided for each patient. The maximum number of patients attending each class will be 12. The classes will combine physical postures (asanas), breathing (pranayama), and deep relaxation (savasana). We would also encourage patient to practice yoga at home and keep a diary.

SUMMARY:
The primary aim of this study is to assess and compare change in QOL during chemotherapy as measured by the Functional Assessment of Cancer Therapy-Breast (FACT-Breast) score between patients receiving yoga and those not receiving yoga. Secondary endpoints will include other measures of QOL such as sleep quality measured with the Pittsburg Sleep Quality Inventory (PSQI), anxiety and depression using Hospital Anxiety and Depression Scale (HADS), and adherence to yoga and to chemotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* History of stage I-III breast cancer
* Patient scheduled to receive or within 2 weeks of receiving intravenous chemotherapy for their breast cancers
* Eastern Cooperative Oncology Group Performance status of <3
* Ability to understand English

5.2 Exclusion Criteria:

* Planning to start yoga on their own within the next 12 weeks
* Maintained a regular personal practice or yoga within the 3 months before enrolling onto the study
* Severe chronic obstructive pulmonary disease
* Class III or IV heart failure
* Child C cirrhosis
* End-Stage renal disease

Exclusion Criteria:

* Planning to start yoga on their own within the next 12 weeks
* Maintained a regular personal practice or yoga within the 3 months before enrolling onto the study
* Severe chronic obstructive pulmonary disease
* Class III or IV heart failure
* Child C cirrhosis
* End-Stage renal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-04; Primary Completion 2018-12-05 (Actual); Study Completion 2018-12-05 (Actual)

PRIMARY OUTCOMES:
change in quality of life | 12 weeks
  to assess and compare change in QOL during chemotherapy as measured by the Functional Assessment of Cancer Therapy-Breast (FACT-Breast) score between patients receiving yoga immediately and those start yoga 3 months later.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Shao, MD, Principal Investigator — Beth Israel Medcial Center
Locations (1):
- Beth Israel Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No